CLINICAL TRIAL: NCT07391059
Title: Randomized Medical Device Class IIa Clinical Investigation to Assess the Safety and Efficacy of a New Shampoo for Head Lice Treatment
Brief Title: Comparative Study for the Evaluation of a New Medical Device Shampoo on the Treatment of Head Lice Infestation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo CSCI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2425CMPH047
Record Dates: First submitted 2025-09-18; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Headlice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INVESTIGATIONAL DEVICE Paranix ® shampoo , 2 MINUTES (Experimental): New medical device shampoo for the treatment of head lice infestation, 2 min treatment time : Paranix ®
  Interventions: Other: INVESTIGATIONAL DEVICE, Paranix ® shampoo 2 minutes
- INVESTIGATIONAL DEVICE Paranix ® shampoo, 5 MINUTES (Experimental): New medical device shampoo for the treatment of head lice infestation, 5 min treatment time : Paranix ®
  Interventions: Other: INVESTIGATIONAL DEVICE, Paranix ® shampoo 5 minutes
- COMPARATOR DEVICE, Pouxit ® shampoo (Active Comparator): Head lice shampoo treatment (medical device class 1) already in market in europe: Pouxit ®
  Interventions: Other: COMPARATOR DEVICE, Pouxit ®

INTERVENTIONS:
Other: INVESTIGATIONAL DEVICE, Paranix ® shampoo 2 minutes — New medical device shampoo for the treatment of head lice infestation: Paranix ® with 2 minute application time
  Arms: INVESTIGATIONAL DEVICE Paranix ® shampoo , 2 MINUTES
Other: INVESTIGATIONAL DEVICE, Paranix ® shampoo 5 minutes — New medical device shampoo for the treatment of head lice infestation: Paranix ®, with 5 minutes application time
  Arms: INVESTIGATIONAL DEVICE Paranix ® shampoo, 5 MINUTES
Other: COMPARATOR DEVICE, Pouxit ® — well established medical device shampoo for the treatment of head lice infestation - Pouxit ®
  Arms: COMPARATOR DEVICE, Pouxit ® shampoo

SUMMARY:
Pediculosis capitis or head lice infestation is a human medical condition caused by the infestation of the hair by the parasitic insect Pediculus humanus capitis (human head lice). The most common symptom of infestation is pruritus (itching) on the head which normally intensifies 3 to 4 weeks after the initial infestation.

The test item has been developed with the ambition to offer a complete head lice treatment, whilst also offering ultimate convenience in use - making treatment of head lice infestation easy, and effective in few minutes.

The objectives of this clinical study are to assess the efficacy and the safety of a new Medical Device shampoo for lice infestation treatment compared to a comparator device, already in market.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant,
* Female or male participants,
* Aged 2 years and above (for participants in arms 1 and 2),
* Aged 3 years and above (for participants in arms 3) ,
* Participants with a slight to moderate lice infestation (According to EU norms: 0, 1, 2)
* Participants with various hair types (from 1 to 3C in the hair scale below) and hair length (from short to mid length hair not exceeding shoulder).
* Written informed consent for participants ≥18 years or legal guardian for participants <18 years given freely and expressly before start of the clinical investigation.
* Participant/Participant's legal guardian is psychologically able to understand the clinical investigation related information and to give written informed consent.
* Participant/participant's legal guardian agreeing to follow the study requirements during the whole clinical investigation period.
* Females of childbearing potential and sexually active should use a contraceptive regimen recognized as effective at least 4 weeks before the beginning of the clinical investigation and during the entire clinical investigation.
* Female participants of childbearing potential, presenting with negative pregnancy test at inclusion.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the clinical investigation;
* Participant who had been deprived of their freedom by an administrative or legal decision or major participant who is under guardianship;
* Participant in a social or sanitary establishment;
* Participant being in an exclusion period from a previous clinical investigation or who is currently participating to another clinical investigation on hair/scalp or who participated to another clinical clinical investigation on hair/scalp within 3 months before first visit.
* Participant suspected to be non-compliant according to the Investigator's judgment.

  * Participant allergic to any of the ingredients and/or materials of the intended to be used products (investigation device and anti-lice comb, comparative device, post-treatment shampoo).

Participant with curly hair (from 4A to 4C in the hair type scale).

* Participant with hair length exceeding shoulder.
* Participants with more than 24 lice on the head.
* Participant suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the clinical investigation results.
* Participant with a cutaneous disease on the studied zone (scalp and hair).
* Severe scratches or open wounds/skin damage on the scalp (lice bites allowed however).
* Participant with a known or suspected allergy to one or more of the components of the investigational or comparator devices.
* Participant who has diabetes.
* Participant with known or suspected immune deficiency or autoimmune disease.

Participant undergoing a topical treatment on the test area or a systemic treatment with:

* anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the clinical investigation;
* corticosteroids during the 2 previous weeks and during the clinical investigation;
* retinoids and/or immunosuppressors during the 3 previous months and during the clinical investigation ;
* any medication stabilized for less than one month.
* Participant who received an anti-lice treatment in the previous month.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Cure Rate after complete treatment | 7 days
  The cure rate is defined as the rate of subjects having no live lice on scalp 7 days after the last application of the product.
Cure Rate after complete treatment | 14 days
  The cure rate is defined as the rate of subjects having no live lice on scalp 7 days after the last application of the product.

SECONDARY OUTCOMES:
Cure rate after one dose of Investigational device (ID) | Day 7
  Comparison of the percentage of participants cured after one dose of the investigational device at 2 minutes compared to the percentage of participants cured with the investigational device at 5 minutes ( after one dose) , compared to the percentage of participants cured with one dose and two doses of the comparator device.
Number of dead and live lice/nymphs after treatment | Day 0 and Day 7 if applicable
  Assessment of the effect of the investigational shampoo on head lice infestation, measured by the number of dead and live lice/nymphs, and the presence of live or unbroken nits collected randomly from the anti-lice comb after treatment. Counting will be done visually using dermatoscope.
Number of live lice and nymphs, after application of treatment | Day 1 and Day 8 if applicable
  Assessment of the effect of the investigational shampoo on head lice infestation, measured by the number of dead and live lice/nymphs, and the presence of live or unbroken nits collected randomly from the anti-lice comb one day after treatment. Counting will be done visually using dermatoscope.
Number of participants with treatment-related adverse events as assessed by investigator | Day 0, Day 1, Day 7, Day 8 and Day 14 if applicable
  Evaluation of the safety and tolerability of the investigational device versus comparator
Subject reported perceived acceptability, effectiveness and subjective evaluation assessed via questionnaire data | Day 1 , Day 7 or Day 14 if applicable
  Evaluation of the perceived acceptability, effectiveness and subjective evaluation. Subject perception questionnaire with:
  * A questionnaire at day 1 consisting of 16 questions with a 4-levels scale (strongly disagree , disagree, agree, strongly agree) and 2 questions with a binary scale (yes, no).
  * A questionnaire at end of study (day 7 or day 14) consisting of 9 questions with a 4-levels scale (strongly disagree , disagree, agree, strongly agree) and 4 questions with a binary scale (yes, no).

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali PETKAR, Dermatologist, Principal Investigator
Locations (1):
- CIDP, Phoenix, Mauritius

IPD SHARING:
Plan to Share IPD: No